CLINICAL TRIAL: NCT02336360
Title: A Multicenter Study to Obtain Data to Assist in Radiation Dosimetry Calculations From Subjects Enrolled in Human Studies Employing 18F-AV-1451
Brief Title: Augmenting Flortaucipir Dosimetry Estimates
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A15
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Urine Analysis (Experimental): Urine will be collected from subjects administered flortaucipir in an Avid-sponsored study to determine the amount of radioactivity excreted in urine.
  Interventions: Drug: Flortaucipir F18

INTERVENTIONS:
Drug: Flortaucipir F18 — No flortaucipir administered in this study. Subjects received flortaucipir in an Avid-sponsored study.
  Other Names: 18F-AV-1451; [F-18]T807; LY3191748; Tauvid

SUMMARY:
This study will obtain data from urine in subjects administered flortaucipir in an Avid-sponsored study to augment the calculation of radiation dosimetry estimates.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who passed screening in an Avid-sponsored study in which flortaucipir will be administered

Exclusion Criteria:

* Subjects who have withdrawn informed consent
* Investigator or sponsor believes it is in the best interest of the subject to be removed from the trials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Molecular NeuroImaging, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred from Jan-Jun 2015 from Avid sponsored study 18F-AV-1451-A05 (NCT02016560)
Groups:
- Urine Analysis: Subjects administered flortaucipir in an Avid-sponsored study consenting to urine radioactivity analysis
Period: Overall Study
Arm/Group | Urine Analysis
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Urine Analysis
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Urine Analysis - Total Integrated Radioactivity Excreted in Urine
Description: Total integrated radioactivity excreted in urine over time will be determined to augment previous radiation dosimetry calculations.
Time Frame: 0-360 minutes post injection
Measure: Mean (Standard Deviation); unit: megabecquerel-hours per megabecquerel
Arm/Group | Urine Analysis
Number analyzed (Participants) | 6
megabecquerel-hours per megabecquerel | 0.1413 (0.07216)

ADVERSE EVENTS:
Time Frame: AEs were not collected in this study
Description: No subjects were administered a drug in this study. Therefore, participants at risk for adverse events in this study is zero.
Arm/Group | Urine Analysis
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less